CLINICAL TRIAL: NCT02493517
Title: A Phase III, Prospective, Randomised, Open Label Study to Compare the Efficacy and Safety of Lanreotide Autogel® 60, 90 or 120 mg With Lanreotide 40 mg PR in Subjects With Active Acromegaly
Brief Title: Efficacy and Safety of Lanreotide Autogel® 60, 90 or 120 mg With Lanreotide 40 mg Prolonged Release (PR) in Acromegaly
Acronym: LANTERN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8-55-52030-289; CTR20140698 (Other: www.ChinaDrugTrials.org.cn)
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lanreotide Autogel® 60mg, 90mg and 120mg (Experimental): Lanreotide Autogel 90mg from day 1 to week 13, 1 injection every 4 weeks (4 in total), titrated to 60mg, 90mg, or 120mg at week 17, then from week 17 to week 29 each group receives 1 injection every 4 weeks (4 in total/group).
  Interventions: Drug: Lanreotide Autogel®
- Lanreotide 40mg PR (Lanreotide Acetate for Injection ) (Active Comparator): Lanreotide PR 40mg from day 1 to week 15, 1 injection every 10 days, then at dose titration (week 16) injection frequency will either remain at 10 days or increase to 14 days or decrease to 7 days up until week 30 or 31.
  Interventions: Drug: Lanreotide Acetate

INTERVENTIONS:
Drug: Lanreotide Autogel® — Lanreotide Autogel 60mg, 90mg, and 120mg, pre-filled syringe, deep subcutaneous injection (provided as a supersaturated solution of lanreotide acetate).
  Arms: Lanreotide Autogel® 60mg, 90mg and 120mg
Drug: Lanreotide Acetate — Lanreotide PR 40mg white freeze-drying cake, 40mg/vial, deep subcutaneous injection (provided as a sterile injectable lyophilisate of lanreotide acetate).
  Arms: Lanreotide 40mg PR (Lanreotide Acetate for Injection )

SUMMARY:
The purpose is to compare the efficacy and safety of lanreotide autogel® 60mg, 90mg or 120mg with lanreotide 40mg PR in subjects with active acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Subject has active acromegaly defined as elevated GH and IGF-1 levels (measured at a central laboratory) as outlined below:

  * A serum level for IGF-1 ≥1.3 x upper limit of normal range (ULN) during the screening period (applicable to both treatment naïve subjects and subjects who have stopped treatment and undergone a washout period prior to Visit 1(Week -4).
  * Subjects must have mean serum GH concentration ≥2.5 μg/L in a GH cycle (5 samples taken at 0, 30, 60, 90 and 120 minutes) during the screening period.
* The subject has undergone surgical removal of an adenoma for acromegaly at least 3 months prior to Screening, or is likely to require pituitary surgery in the future but not before completing at least 32 weeks of study treatment plus an additional follow up of 8 weeks for subjects taking part in the pharmacokinetics (PK) extension, or for whom pituitary surgery is not an option (due to contraindications, refusal etc.) and is therefore never likely to undergo pituitary surgery.

Exclusion Criteria:

* The subject has been treated with radiotherapy within 10 years prior to Screening.
* The subject has been treated with lanreotide Autogel, lanreotide PR, pegvisomant, cabergoline or octreotide LAR within 3 months of Screening or octreotide immediate release (IR) or bromocriptin within 2 weeks of Screening.
* The subject has a history of or currently presents with clinically significant ventricular or atrial dysrhythmias ≥Grade 2, using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0.
* The subject has uncontrolled diabetes (glycosylated haemoglobin (HbA1c) >8.5%).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- China (10):
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Provincial Hospital, Fuzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Affiliate Hospital of Guiyang Medical College, Guizhou
  - Jiangsu Provincial People's Hospital, Nanjing
  - Huashan Hospital Fudan University, Shanghai
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Medical College Huazhong University of Science & Technology, Wuhan

REFERENCES:
- [Derived] An Z, Lei T, Duan L, Hu P, Gou Z, Zhang L, Durand-Gasselin L, Wang N, Wang Y, Gu F; LANTERN study investigators. Efficacy and safety of lanreotide autogel compared with lanreotide 40 mg prolonged release in Chinese patients with active acromegaly: results from a phase 3, prospective, randomized, and open-label study (LANTERN). BMC Endocr Disord. 2020 May 4;20(1):57. doi: 10.1186/s12902-020-0524-7. PMID 32366244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult subjects with active acromegaly, defined as elevated Insulin-like Growth Factor 1 (IGF-1) and Growth Hormone (GH) levels, were recruited into 10 study sites in China.
Pre-assignment Details: 170 subjects were screened and 128 eligible subjects were stratified according to surgical history (previous pituitary surgery or no previous pituitary surgery) and randomised in a 1:1 ratio to receive lanreotide Autogel or lanreotide prolonged release (PR). All randomised subjects were treated.
Groups:
- Lanreotide Autogel: Subjects were randomised to receive lanreotide Autogel. Lanreotide Autogel was administered subcutaneously (s.c.) at a fixed dose of 90 milligrams (mg) every 4 weeks from Day 1, Week 1 to Week 17. At Week 17 the dose was continued at 90 mg or titrated to 60 mg or 120 mg, administered every 4 weeks according to the individual subject's response as determined by the mean value of the GH cycles and IGF-1 measured at the previous Week 13 Visit. The last dose of lanreotide Autogel was given at Week 29, followed by End of Study Treatment (EOST) / Early Withdrawal (EW) Visit at Week 33.
- Lanreotide PR: Subjects were randomised to receive lanreotide PR. Lanreotide PR was administered intramuscularly (i.m.) every 10 days from Day 1, Week 1 up to Week 16. At Week 16 the injection interval was maintained at 10 days or was adjusted to 7 or 14 days according to the individual subject's response as determined by the mean value of GH cycle and IGF-1 measured at the previous Week 13 Visit. The last dose of lanreotide PR was administered at Week 31. The EOST/EW Visit was at Week 32.
Period: Overall Study
Arm/Group | Lanreotide Autogel | Lanreotide PR
Started | 64 | 64
Completed | 62 | 57
Not Completed | 2 | 7
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Missed study visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the Safety population which consisted of all randomised subjects who received at least one dose of study treatment. The Safety population was analysed using subjects as treated.
Groups:
- Lanreotide Autogel: Subjects were randomised to receive lanreotide Autogel. Lanreotide Autogel was administered s.c. at a fixed dose of 90 mg every 4 weeks from Day 1, Week 1 to Week 17. At Week 17 the dose was continued at 90 mg or titrated to 60 mg or 120 mg every 4 weeks according to the individual subject's response as determined by the mean value of the GH cycles and IGF-1 measured at the previous Week 13 Visit. The last dose of lanreotide Autogel was given at Week 29, followed by EOST/EW Visit at Week 33.
- Lanreotide PR: Subjects were randomised to receive lanreotide PR. Lanreotide PR was administered i.m. every 10 days from Day 1, Week 1 up to Week 16. At Week 16 the injection interval was maintained at 10 days or was adjusted to 7 or 14 days according to the individual subject's response as determined by the mean value of GH cycle and IGF-1 measured at the previous visit at Week 13. The last dose of lanreotide PR was administered at Week 31. The EOST/EW Visit was at Week 32.
Arm/Group | Lanreotide Autogel | Lanreotide PR | Total Title
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (11.2) | 40.8 (12.6) | 39.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 26 | 24 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 64 | 64 | 128
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Standardised Mean Change From Baseline in Age-adjusted IGF-1 Levels at the EOST/EW Visit
Description: The standardised mean change from Baseline in age-adjusted log-transformed IGF-1 standard deviation score (SDS) at EOST/EW is presented for subjects treated with both lanreotide Autogel and lanreotide PR. Back-transformed results are presented in addition to the results without back-transformation.
  For each subject the IGF-1 SDS value was calculated based on the z-score derivation: IGF-1 SDS = (IGF-1 - mean)/ standard deviation (SD), with mean and SD derived from the upper limit of normal (ULN) and lower limit of normal (LLN) margins for each age category. ULN = Mean + 2 SD; LLN = Mean - 2 SD.
  The SDS indicates the number of standard deviations away from the mean. A SDS of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. A negative change in the SDS indicates a decrease in the mean age-adjusted IGF-1 values.
Time Frame: Baseline to EOST/EW Visit (up to Week 33 for the lanreotide Autogel group and up to Week 32 for the lanreotide PR group).
Population: The Per Protocol population consisted of all subjects who were randomised and treated with at least one baseline and at least one postbaseline assessment of the primary efficacy parameter and for whom no major protocol deviations occurred with impact on efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: SDS
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 54 | 44
SDS
  Without back-transformation | -0.84 (0.15) | -0.52 (0.17)
  With back transformation | 0.43 (1.16) | 0.59 (1.19)
Statistical Analysis 1: Comparison: Lanreotide Autogel vs Lanreotide PR; The Least Square (LS) Means and 95% Confidence Intervals (CIs) were based on the generalised linear model (GLM) with IGF-1 SDS change from baseline values as dependent variable, with treatment group and previous pituitary surgery as independent factors, and the baseline value of IGF-1 SDS as independent covariate. A log-transformation with base e was applied to the IGF-1 SDS data before analysing. The treatment difference (lanreotide Autogel - lanreotide PR) is presented; Test type: Non-Inferiority — The non-inferiority margin is defined as 0.6 SDS for the upper limit of 95% CI of the LS mean difference of the log-transformed IGF-1 SDS without back-transformation; Treatment difference = -0.32, 95% CI 2-sided [-0.74 to 0.11]
Statistical Analysis 2: Comparison: Lanreotide Autogel vs Lanreotide PR; The LS Means and 95% CIs were based on the GLM with IGF-1 SDS change from baseline values as dependent variable, with treatment group and previous pituitary surgery as independent factors, and the baseline value of IGF-1 SDS as independent covariate. A log-transformation with base e was applied to the IGF-1 SDS data before analysing. The LS Mean ratio (lanreotide Autogel versus lanreotide PR) is presented; Test type: Non-Inferiority — The non-inferiority margin for the back-transformed LS Mean ratio of IGF-1 SDS of lanreotide Autogel versus lanreotide PR is exp (0.6) = 1.822; LS Mean ratio = 0.73, 95% CI 2-sided [0.48 to 1.11]

2. Secondary Outcome: Percentage of Subjects With Normal Age-adjusted IGF-1 Levels at the EOST/EW Visit
Description: The percentage of subjects with normal age-adjusted IGF-1 levels at the EOST/EW Visit is presented for subjects treated with Lanreotide Autogel and Lanreotide PR.
  At baseline, all subjects had abnormal IGF-1 levels as per protocol entry criteria.
Time Frame: as for outcome 1
Population: The Intention-To-Treat (ITT) population consisted of all randomised and treated subjects who had at least one baseline and at least one postbaseline assessment of the primary efficacy parameter. The ITT population was analysed using subjects as randomised.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 64 | 64
Percentage of Subjects | 15.6 | 9.4
Statistical Analysis 1: Comparison: Lanreotide Autogel vs Lanreotide PR; The risk difference (lanreotide Autogel - lanreotide PR) in the percentage of normal IGF-1 SDS values at EOST/EW Visit is presented; Test type: Other; Risk Difference (RD) = 6.3, 95% CI 2-sided [-5.2 to 17.7]

3. Secondary Outcome: Percentage of Subjects With GH ≤2.5 Micrograms Per Litre (mcg/L) at the EOST/EW Visit
Description: The percentage of subjects with GH ≤2.5 mcg/L at the EOST/EW Visit is presented for subjects treated with lanreotide Autogel and lanreotide PR.
  At baseline, all subjects had GH levels >2.5 mcg/L as per protocol entry criteria.
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomised and treated subjects who had at least one baseline and at least one postbaseline assessment of the primary efficacy parameter. The ITT population was analysed using subjects as randomised.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 64 | 64
Percentage of Subjects | 29.7 | 31.3
Statistical Analysis 1: Comparison: Lanreotide Autogel vs Lanreotide PR; The risk difference (lanreotide Autogel - lanreotide PR) in the percentage of GH levels ≤2.5 mcg/L at EOST/EW Visit is presented; Test type: Other; Risk Difference (RD) = -1.6, 95% CI 2-sided [-17.5 to 14.4]

4. Secondary Outcome: The Percentage of Subjects With GH ≤1 mcg/L at the EOST/EW Visit
Description: The percentage of subjects with GH ≤1 mcg/L at the EOST/EW Visit is presented for subjects treated with lanreotide Autogel and lanreotide PR.
  At baseline, all subjects had GH levels >2.5 mcg/L as per protocol entry criteria.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Percentage of Subjects
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 64 | 64
Percentage of Subjects | 10.9 | 9.4
Statistical Analysis 1: Comparison: Lanreotide Autogel vs Lanreotide PR; The risk difference (lanreotide Autogel - lanreotide PR) in the percentage of GH levels ≤1 mcg/L at EOST/EW Visit is presented; Test type: Other; Risk Difference (RD) = 1.6, 95% CI 2-sided [-8.9 to 12.0]

5. Secondary Outcome: Percentage of Subjects With Normal Age-adjusted IGF-1 Levels and Who Have GH Levels >1 mcg/L and ≤2.5 mcg/L at the EOST/EW Visit
Description: The percentage of subjects with normal age-adjusted IGF-1 levels and who have GH levels >1 mcg/L but ≤2.5 mcg/L at the EOST/EW Visit is presented for subjects treated with lanreotide Autogel and lanreotide PR. The calculation of percentages was based on the overall ITT population.
  At baseline, all subjects had abnormal IGF-1 levels and GH levels >2.5 mcg/L as per protocol entry criteria.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number; unit: Percentage of Subjects
Groups:
- Lanreotide PR: Subjects were randomised to receive lanreotide PR. Lanreotide PR was adminsitered i.m. every 10 days from Day 1, Week 1 up to Week 16. At Week 16 the injection interval was maintained at 10 days or was adjusted to 7 or 14 days according to the individual subject's response as determined by the mean value of GH cycle and IGF-1 measured at the previous visit at Week 13. The last dose of lanreotide PR was administered at Week 31. The EOST/EW Visit was at Week 32.
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 64 | 64
Percentage of Subjects | 7.8 | 3.1
Statistical Analysis 1: Comparison: Lanreotide Autogel vs Lanreotide PR; The risk difference (lanreotide Autogel - lanreotide PR) in the percentage subjects with normal IGF-1 levels and who have GH levels >1 mcg/L and ≤2.5 mcg/L at EOST/EW Visit is presented; Test type: Other; Risk Difference (RD) = 4.7, 95% CI 2-sided [-3.1 to 12.5]

6. Secondary Outcome: Mean Change From Baseline in GH Values at the EOST/EW Visit
Description: The mean change from baseline in GH values at the EOST/EW Visit is presented for subjects treated with lanreotide Autogel and lanreotide PR.
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomised and treated subjects who had at least one baseline and at least one postbaseline assessment of the primary efficacy parameter. The ITT population was analysed using subjects as randomised. Subjects with data available at time of analysis are presented.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 64 | 62
mcg/L | -9.548 (22.852) | -13.182 (20.224)
Statistical Analysis 1: Comparison: Lanreotide Autogel vs Lanreotide PR; Treatment difference (lanreotide Autogel - lanreotide PR) is presented; Test type: Other; Treatment difference = 3.63, 95% CI 2-sided [-3.98 to 11.25], Standard Deviation 21.60

7. Secondary Outcome: Percentage of Subjects With at Least 20% Reduction in Tumour Volume at EOST/EW Visit Compared to Baseline
Description: The percentage of subjects with at least a 20% reduction in the solid component of the tumour volume at the EOST/EW Visit compared to baseline is presented for the subgroup of subjects who had solid tumours at baseline.
  The tumour volume was measured by Magnetic Resonance Imaging (MRI) at Screening and at the EOST/EW Visit, and then assessed by two independent blinded readers.
Time Frame: as for outcome 1
Population: The ITT population consisted of all randomised and treated subjects who had at least one baseline and at least one postbaseline assessment of the primary efficacy parameter. The ITT population was analysed using subjects as randomised. Data is presented for the subgroup of subjects in the ITT population who had solid tumours at baseline.
Measure: Number; unit: Percentage of Subjects
Groups:
- Lanreotide PR: Subjects were randomised to receive lanreotide PR. Lanreotide PR was administered i.m.every 10 days from Day 1, Week 1 up to Week 16. At Week 16 the injection interval was maintained at 10 days or was adjusted to 7 or 14 days according to the individual subject's response as determined by the mean value of GH cycle and IGF-1 measured at the previous visit at Week 13. The last dose of lanreotide PR was administered at Week 31. The EOST/EW Visit was at Week 32.
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 55 | 53
Percentage of Subjects | 45.5 | 50.9
Statistical Analysis 1: Comparison: Lanreotide Autogel vs Lanreotide PR; Risk difference (lanreotide Autogel - lanreotide PR) in the percentage of subjects with at least 20% reduction in the solid component of tumour volume compared to Baseline is presented; Test type: Other; Risk Difference (RD) = -5.5, 95% CI 2-sided [-24.3 to 13.3]

8. Secondary Outcome: Median Percentage Change From Baseline in Tumour Volume at the EOST/EW Visit
Description: The median percentage change in the solid component of the tumour volume from baseline to the EOST/EW Visit is presented.
  The tumour volume was measured by MRI at Screening and at the EOST/EW Visit, and then assessed by two independent blinded readers.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Median (Full Range); unit: Percentage change in tumour volume
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 55 | 53
Percentage change in tumour volume | -17.870 [-75.77 to 95259.11] | -20.120 [-86.41 to 113.03]

9. Secondary Outcome: Percentage of Subjects With at Least One Symptom of Acromegaly at Week 13 and at the EOST/EW Visit Compared to Baseline
Description: The percentage of subjects with at least one symptom of acromegaly at Week 13 and at the EOST/EW Visit compared with baseline is presented for subjects treated with lanreotide Autogel and lanreotide PR. The symptoms of acromegaly monitored included: headache, excessive perspiration, fatigue, soft tissue swelling and arthralgia.
Time Frame: Baseline, Week 13 Visit and EOST/EW Visit (up to Week 33 for the lanreotide Autogel group and up to Week 32 for the lanreotide PR group).
Population: as for outcome 3
Measure: Number; unit: Percentage of Subjects
Arm/Group | Lanreotide Autogel | Lanreotide PR
Number analyzed (Participants) | 64 | 64
Percentage of Subjects
  Week 13 Visit | 70.3 | 59.4
  EOST/EW Visit | 75.0 | 59.4

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from the first dose of study treatment up to the EOST/EW Visit (up to approximately 33 weeks).
Description: TEAEs were reported for the Safety population which consisted of all randomised subjects who received at least one dose of study treatment. The Safety population was analysed using subjects as treated.
Arm/Group | Lanreotide Autogel | Lanreotide PR
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/64 | 2/64
Other Adverse Events (participants affected / at risk) | 59/64 | 62/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel (N=64) | Lanreotide PR (N=64)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel (N=64) | Lanreotide PR (N=64)
Diarrhoea (Gastrointestinal disorders) | 51 (194) | 46 (337)
Abdominal distension (Gastrointestinal disorders) | 22 (67) | 27 (146)
Abdominal pain (Gastrointestinal disorders) | 18 (40) | 20 (114)
Abdominal pain upper (Gastrointestinal disorders) | 13 (32) | 16 (37)
Nausea (Gastrointestinal disorders) | 7 (7) | 16 (69)
Constipation (Gastrointestinal disorders) | 7 (14) | 10 (14)
Flatulence (Gastrointestinal disorders) | 7 (8) | 3 (5)
Toothache (Gastrointestinal disorders) | 4 (4) | 5 (8)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 3 (5)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 3 (7) | 9 (32)
Gastric dilatation (Gastrointestinal disorders) | 2 (2) | 4 (7)
Rectal tenesmus (Gastrointestinal disorders) | 1 (1) | 9 (37)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (9)
Cholelithiasis (Hepatobiliary disorders) | 23 (27) | 18 (19)
Gallbladder enlargement (Hepatobiliary disorders) | 4 (4) | 3 (3)
Cholestasis (Hepatobiliary disorders) | 4 (4) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 3 (3) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 21 (28) | 18 (31)
Nasopharyngitis (Infections and infestations) | 7 (17) | 10 (12)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (2)
Weight decreased (Investigations) | 8 (9) | 4 (4)
Blood glucose increased (Investigations) | 7 (7) | 6 (6)
Protein urine present (Investigations) | 3 (3) | 4 (4)
Blood parathyroid hormone increased (Investigations) | 1 (1) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (12) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 10 (15) | 0 (0)
Injection site induration (General disorders) | 6 (8) | 14 (33)
Chest discomfort (General disorders) | 3 (9) | 5 (10)
Pyrexia (General disorders) | 3 (4) | 4 (4)
Injection site pain (General disorders) | 2 (2) | 9 (38)
Injection site swelling (General disorders) | 0 (0) | 6 (24)
Headache (Nervous system disorders) | 10 (17) | 17 (61)
Dizziness (Nervous system disorders) | 6 (11) | 10 (19)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (8)
Renal cyst (Renal and urinary disorders) | 4 (4) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 3 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Sinus bradycardia (Cardiac disorders) | 9 (9) | 12 (12)
Thyroid mass (Endocrine disorders) | 4 (4) | 7 (7)
Hypothyroidism (Endocrine disorders) | 1 (1) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Hypertension (Vascular disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other